CLINICAL TRIAL: NCT03702881
Title: Anterior Open Bite Treatment With Bonded Spurs Associated With Build-ups Versus Conventional Bonded Spurs: a Randomized Clinical Trial.
Brief Title: Anterior Open Bite Treatment With Bonded Spurs Associated With Build-ups Versus Conventional Bonded Spurs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Aron Aliaga-Del Castillo, DDS, MSc., PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68551617.8.0000.5417
Record Dates: First submitted 2018-10-07; First posted 2018-10-11 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Malocclusion; Open Bite
Keywords: Open Bite; Orthodontic appliance; Cephalometry; Dental models
MeSH Terms: conditions — Malocclusion; Open Bite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bonded Spurs associated with posterior build-ups Group (Experimental): The experimental group will consist of 25 patients treated with bonded spurs associated with build-ups.
  Interventions: Device: Bonded Spurs associated with posterior build-ups
- Conventional bonded spurs Group (Active Comparator): Active comparator group will consist of 25 patients treated with conventional bonded spurs
  Interventions: Device: Conventional bonded spurs

INTERVENTIONS:
Device: Bonded Spurs associated with posterior build-ups — Twenty-five patients will be treated with bonded spurs associated with posterior build-ups. The cervical portion of the palatal surfaces of the maxillary incisors and the incisal portion of the lingual surfaces of the mandibular incisors will be pumiced, rinsed, dried, and acid etched with 37% phosphoric acid. The etched surfaces will be subsequently rinsed and carefully dried. Then, the spurs will be bonded using Transbond primer/adhesive. The positions for the spurs will be chose to prevent possible future occlusal interferences The spurs will be sharpened with a carborundum disk before bonding. In addition, posterior build-ups (resin blocks) will be cemented on the functional cusps of all maxillary posterior teeth. The treatment time will be 12 months. After this time, the posterior build ups will be removed and the bonded spurs will be maintained for 12 months more, as active retention.
  Arms: Bonded Spurs associated with posterior build-ups Group
Device: Conventional bonded spurs — Twenty-five patients will be treated only with bonded spurs. The bonding of the spurs will follow the same protocol described for the experimental group. The treatment time will be 12 months. After this time, the bonded spurs will be maintained for 12 months more, as active retention.
  Arms: Conventional bonded spurs Group

SUMMARY:
This study compares the dentoalveolar and skeletal effects of bonded spurs associated with build-ups versus conventional bonded spurs in the early treatment of anterior open bite patients. Half of participants will be treated with bonded spurs associated with build-ups, while the other half will be treated with conventional bonded spurs.

The null hypothesis to be tested is that there are no differences for the dentoalveolar and skeletal effects between the two protocols.

DETAILED DESCRIPTION:
Anterior open bite is commonly related with lower anterior face height increase. Some early treatment protocols use appliances that control deleterious habits associated to appliances that produce control of the vertical dimension. Usually, these appliances (chincup, removable orthopedics) depend on patient's collaboration. Recently, the efficiency and stability of anterior open bite treatment with resin blocks bonded to the posterior teeth (build-ups) associated with fixed orthodontic appliances was described. They could be considered as a promissory alternative for vertical control during anterior open bite treatment. Then, it could be thought that the association of bonded spurs with posterior build-ups, instead of chincup, would produce vertical control during anterior open bite early treatment without the need of patient collaboration. Therefore, the aim of this study is to compare the dentoalveolar and skeletal effects of bonded spurs associated with build-ups versus conventional bonded spurs in the early treatment of anterior open bite patients.

For this, patients will be recruited at the Orthodontic Clinic of Bauru Dental School, University of São Paulo, Brazil. Fifty patients between 7 and 11 years old diagnosed with anterior open bite greater than 1 mm will be prospective and randomly allocated in one of the two study group. The experimental group will consist of 25 patients treated with bonded spurs associated with build-ups. Control group will consist of 25 patients treated with conventional bonded spurs.

Lateral radiographs and digital dental models will be obtained at the beginning (T1), 12 months after treatment (T2), and 24 months after treatment (T3). Dentoalveolar and skeletal variables will be evaluated from the lateral radiographs in the Dolphin® software. Dental casts will be analyzed with the Orthoanalyzer® software to evaluate dentoalveolar anterior vertical development, posterior teeth inclinations and arch dimensions. Superimposition of digital dental models will be performed to evaluate the relative three-dimensional dentoalveolar changes on the maxillary and mandibular arches. Discomfort, pain and quality of life will be evaluated using questionnaires.

After verifying the normal distribution, intergroup comparisons (T1 vs T2 and T1 vs T3) will be performed with t test and intragroup comparisons with dependent t test. Results will be considered statistically significant at P<0.05.

The possible harms that could appear with these therapies are related to temporary tongue discomfort during the first days after the installation of the appliances. Patients and parents will be informed that is it normal. Although it has been reported that the discomfort is temporary and transitory and usually patients adapted to the treatment after 3-5 days, patients or parents will be able to stop the treatment at any moment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 7 to 11 years old,
* erupted permanent first permanent molars,
* anterior open bite (AOB) greater than 1 mm,
* maxillary and mandibular permanent central incisors fully erupted,
* no or mild crowding,
* without the need of maxillary expansion
* Children in the first transitional period will be considered to be eligible for treatment when the maxillary lateral incisors are beginning to erupt and the maxillary central incisors still show an open bite

Exclusion Criteria:

* previous orthodontic treatment,
* craniofacial anomalies or syndromes,
* tooth agenesis,
* loss of permanent teeth,
* severe crowding,
* maxillary constriction or posterior crossbite

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Overbite (mm) | 12 months
Gonial angle (º) | 12 months
Mandibular plane angle (º) | 12 months
Maxillary and mandibular molar vertical development (mm) | 12 months

SECONDARY OUTCOMES:
Overbite (mm) | 24 months
Gonial angle (º) | 24 months
Mandibular plane angle (º) | 24 months
Maxillary and mandibular molar vertical development (mm) | 24 months
Maxillary and mandibular position (º) | 12 months
Maxillary and mandibular position (º) | 24 months
Maxillary and mandibular length (mm) | 12 months
Maxillary and mandibular length (mm) | 24 months
Mandibular ramus height (mm) | 12 months
Mandibular ramus height (mm) | 24 months
Sagittal skeletal discrepancy (º) | 12 months
Sagittal skeletal discrepancy (º) | 24 months
Facial axis angle (º) | 12 months
Facial axis angle (º) | 24 months
Maxillomandibular divergence angle (º) | 12 months
Maxillomandibular divergence angle (º) | 24 months
Palatal plane inclination (º) | 12 months
Palatal plane inclination (º) | 24 months
Anterior face height (mm) | 12 months
Anterior face height (mm) | 24 months
Posterior face height (mm) | 12 months
Posterior face height (mm) | 24 months
Lower anterior face height (mm) | 12 months
Lower anterior face height (mm) | 24 months
Overjet (mm) | 12 months
Overjet (mm) | 24 months
Maxillary and mandibular incisors Inclination (º) | 12 months
Maxillary and mandibular incisors Inclination (º) | 24 months
Maxillary and mandibular incisors position (mm) | 12 months
Maxillary and mandibular incisors position (mm) | 24 months
Maxillary and mandibular incisors height (mm) | 12 months
Maxillary and mandibular incisors height (mm) | 24 months
Nasolabial angle (º) | 12 months
Nasolabial angle (º) | 24 months
Upper lip inclination (º) | 12 months
Upper lip inclination (º) | 24 months
Upper and lower lip position (mm) | 12 months
Upper and lower lip position (mm) | 24 months
Interlabial gap (mm) | 12 months
Interlabial gap (mm) | 24 months
Maxillary and mandibular anterior dentoalveolar vertical development (mm) | 12 months
Maxillary and mandibular anterior dentoalveolar vertical development (mm) | 24 months
Bucco-lingual inclinations of maxillary and mandibular permanent first molars (º) | 12 months
Bucco-lingual inclinations of maxillary and mandibular permanent first molars (º) | 24 months
Maxillary and mandibular inter-first permanent molar distances (mm) | 12 months
Maxillary and mandibular inter-first permanent molar distances (mm) | 24 months
Maxillary and mandibular inter-canine distances (mm) | 12 months
Maxillary and mandibular inter-canine distances (mm) | 24 months
Maxillary and mandibular arch perimeters (mm) | 12 months
Maxillary and mandibular arch perimeters (mm) | 24 months
Maxillary and mandibular arch lengths (mm) | 12 months
Maxillary and mandibular arch lengths (mm) | 24 months
Palatal depth (mm) | 12 months
Palatal depth (mm) | 24 months
Dentoalveolar displacements obtained from three-dimensional superimposition (mm) | 12 months
Dentoalveolar displacements obtained from three-dimensional superimposition (mm) | 24 months
Discomfort and pain intensity evaluated with questionnaires | 1 month
  A 10-cm Visual Analog Scale will be used, where "0-cm" is the minimum score indicating nor discomfort or pain intensity and "10-cm" is the maximum score denoting the greatest discomfort or pain intensity.
Discomfort and pain intensity evaluated with questionnaires | 12 months
  A 10-cm Visual Analog Scale will be used, where "0-cm" is the minimum score indicating nor discomfort or pain intensity and "10-cm" is the maximum score denoting the greatest discomfort or pain intensity.
Discomfort and pain intensity evaluated with questionnaires | 24 months
  A 10-cm Visual Analog Scale will be used, where "0-cm" is the minimum score indicating nor discomfort or pain intensity and "10-cm" is the maximum score denoting the greatest discomfort or pain intensity.
Parent´s perception of children discomfort and pain intensity evaluated with questionnaires | 1 month
  A 10-cm Visual Analog Scale will be used, where "0-cm" is the minimum score indicating nor discomfort or pain intensity and "10-cm" is the maximum score denoting the greatest discomfort or pain intensity.
Quality of life evaluation with questionnaires | 12 months
  Oral health related-quality of life evaluation will be performed with the Child Perceptions Questionnaire (CPQ8-10). The questionnaire contains 25 items distributed in four domains: oral symptoms, functional limitations, emotional wellbeing and social wellbeing. The items assess the frequency of the events that occurs in the four weeks previous to the application of the questionnaire. A 5-point Likert scale is used with the options: Never (0), Once/twice (1), Sometimes (2), Often (3), and Every day/almost every day (4). The CPQ8-10 scores are obtained by summing all item scores. The total score ranges from "0" indicating no impact of oral condition on quality of life, to "100" indicating maximal impact of oral condition on quality of life.
Quality of life evaluation with questionnaires | 24 months
  Oral health related-quality of life evaluation will be performed with the Child Perceptions Questionnaire (CPQ8-10). The questionnaire contains 25 items distributed in four domains: oral symptoms, functional limitations, emotional wellbeing and social wellbeing. The items assess the frequency of the events that occurs in the four weeks previous to the application of the questionnaire. A 5-point Likert scale is used with the options: Never (0), Once/twice (1), Sometimes (2), Often (3), and Every day/almost every day (4). The CPQ8-10 scores are obtained by summing all item scores. The total score ranges from "0" indicating no impact of oral condition on quality of life, to "100" indicating maximal impact of oral condition on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru Dental School, University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aliaga-Del Castillo A, Maranon-Vasquez GA, Janson G, Vilanova L, Miranda F, Massaro C, Bellini-Pereira SA, Arriola-Guillen LE, Yatabe M, Ruellas AC, Cevidanes L, Garib D. Oral health-related quality of life, adaptation/discomfort during open bite treatment with spurs: complementary analysis from a randomized clinical trial. Sci Rep. 2024 Mar 8;14(1):5732. doi: 10.1038/s41598-024-56363-0. PMID 38459254
- [Derived] Aliaga-Del Castillo A, Janson G, Vilanova L, Cevidanes L, Yatabe M, Garib D, Arriola-Guillen LE, Miranda F, Massaro C, Bellini-Pereira SA, Ruellas AC. Three-dimensional dentoalveolar changes in open bite treatment in mixed dentition, spurs/posterior build-ups versus spurs alone: 1-year follow-up randomized clinical trial. Sci Rep. 2022 Jul 20;12(1):12378. doi: 10.1038/s41598-022-15988-9. PMID 35858941
- [Derived] Aliaga-Del Castillo A, Bellini-Pereira SA, Vilanova L, Miranda F, Massaro C, Arriola-Guillen LE, Garib D, Janson G. Dental arch changes after open bite treatment with spurs associated with posterior build-ups in the mixed dentition: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2021 Jun;159(6):714-723.e1. doi: 10.1016/j.ajodo.2020.11.036. Epub 2021 Mar 30. PMID 33795189
- [Derived] Aliaga-Del Castillo A, Vilanova L, Miranda F, Arriola-Guillen LE, Garib D, Janson G. Dentoskeletal changes in open bite treatment using spurs and posterior build-ups: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2021 Jan;159(1):10-20. doi: 10.1016/j.ajodo.2020.06.031. Epub 2020 Nov 18. PMID 33221096